CLINICAL TRIAL: NCT02575001
Title: The Influence of Psychobiological Adversity to Children and Adolescents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Attachment2015
Record Dates: First submitted 2015-07-23; First posted 2015-10-14 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes; Stress
Keywords: Type 1 diabetes; Children and adolescents; Stress; Genetic factors; Psychological background
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The genes with expected influence to stress reactivity and mental disorders will be tested.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 diabetes: Children with Type 1 diabetes, age from 8 to 15 years.
  The following interventions/exposures will be administered:
  Behavioral: Psychological background determinations, Genetic: Genetic susceptibility determination, Procedure/Surgery: Cortisol release test, Procedure/Surgery: Saliva cortisol measurement.
  Interventions: Behavioral: Psychological background determinations; Genetic: Genetic susceptibility determination; Procedure: Cortisol release test; Procedure: Saliva cortisol measurement
- Healthy control: Healthy primary school pupils, age from 8 to 15 years.
  The following interventions/exposures will be administered:
  Behavioral: Psychological background determinations, Genetic: Genetic susceptibility determination, Procedure/Surgery: Saliva cortisol measurement.
  Interventions: Behavioral: Psychological background determinations; Genetic: Genetic susceptibility determination; Procedure: Saliva cortisol measurement

INTERVENTIONS:
Behavioral: Psychological background determinations — For the psychological background determinations a structured interview and questionnaires will be administered:
  1. Child Attachment Interview (CAI)
  2. General/sociodemographic questionnaire with the questions on diabetes management, current health status and the child's development in the infancy
  3. "Parenting Stress Index" with the "19-item Life Stress Scale" (PSI)
  4. Achenbach System of Empirically Based Assessment (CBCL, YSR)
  5. Holmes and Rahe "Social readjustment rating scale"
  6. Lifetime Incidence of Traumatic Events (LITE) - parent and child reports of child's trauma/loss history (LITE- S/ P)
  7. Experiences in Close Relationships - Relationship Structures questionnaire (ECR-RS)
Genetic: Genetic susceptibility determination — DNA will be isolated from the patients' blood samples and form the control subjects buccal swabs. The genes with expected influence to stress reactivity and mental disorders will be tested.
Procedure: Cortisol release test — Synacthen test - will be used with the group of patients with type 1 diabetes to measure HPA axis reactivity
  Groups: Type 1 diabetes
Procedure: Saliva cortisol measurement — Saliva cortisol measurement - will be used with the patients before and after the Synacthen test and with the Hashimoto thyroiditis and the healthy control group before and after the Child Attachment Interview

SUMMARY:
The aims of this study are two fold: To show whether there is an increased environmental or genetic susceptibility to stress in patients with T1D and whether it influences diabetes management. And to develop a strategy for the assessment and treatment of patients with T1D and an increased risk for development of psychopathology under stress.

DETAILED DESCRIPTION:
Lately, a marked increase in the incidence and earlier age of onset of type 1 diabetes (T1D) has been noted. These observations could also be connected to an increased prevalence of stressful experiences and a lowered stress tolerance in some children.

The way a person responds to stress is determined by the interplay of genetic and environmental factors. Environmental experiences at specific times of development have been shown to shape individual's hypothalamic-pituitary-adrenal axis (HPA axis) stress response. It is known, that early development of central nervous system is critically dependent on child's interaction with the environment (experience dependent maturation), especially to the attachment to caregivers (most often the mother). Appropriate caregiving is connected to lower basal cortisol levels in children and a more stable HPA axis response after the exposure to stress. Any circumstances that disturbed the formation of the attachment to the primary caregiver (e.g. complications at delivery, psychosocial stressors affecting the mother or mother's postpartum depression) resulted in higher HPA axis responsiveness to stress in the affected children.

Changes in individual genes have also been shown to influence a person's susceptibility to stress and risk for the development of stress-induced psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by a parent/legal guardian and informed assent signed by the study participant prior study entry
* Diagnosed with Type 1 DM prior to signature of Patient Informed Consent (PIC) (for the T1D group).
* Age between 8-15 years old (inclusive) at signature of PIC
* Treated by the investigator's centre prior signature of PIC (For the T1D group).
* Willing to undergo all study procedures

Exclusion Criteria:

* Any documented concomitant chronic disease known to affect diabetes control (e.g. altered renal function, active cancer undergoing treatment, Crohn's disease, ulcerative colitis, Mb Addison disease)
* Any other medical, social or psychological condition that, in the investigator's opinion, makes the patient unable to comply with the study protocol (e.g. intellectual disability).

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children of 8 to 15 years of age with type 1 diabetes with their parents; Healthy primary school pupils of 8 to 15 years of age with their parents
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Significant between group differences in metabolic control | 1 month
  Association between psychological scores, stress reactivity, genetic factors and metabolic control in patients with type 1 diabetes

SECONDARY OUTCOMES:
Significant differences in psychological scores between groups | 1 week
  Significant differences in psychological scores between the patients with type 1 diabetes and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, MD, PhD, Principal Investigator — University of Ljubljana, Faculty of Medicine
Locations (1):
- University of Ljubljana, Faculty of Medicine, Ljubljana, Slovenia

REFERENCES:
- [Background] Nolte T, Guiney J, Fonagy P, Mayes LC, Luyten P. Interpersonal stress regulation and the development of anxiety disorders: an attachment-based developmental framework. Front Behav Neurosci. 2011 Sep 21;5:55. doi: 10.3389/fnbeh.2011.00055. eCollection 2011. PMID 21960962
- [Background] Lupien SJ, Fiocco A, Wan N, Maheu F, Lord C, Schramek T, Tu MT. Stress hormones and human memory function across the lifespan. Psychoneuroendocrinology. 2005 Apr;30(3):225-42. doi: 10.1016/j.psyneuen.2004.08.003. PMID 15511597
- [Background] McEwen BS. Protective and damaging effects of stress mediators. N Engl J Med. 1998 Jan 15;338(3):171-9. doi: 10.1056/NEJM199801153380307. No abstract available. PMID 9428819
- [Background] McEwen BS, Biron CA, Brunson KW, Bulloch K, Chambers WH, Dhabhar FS, Goldfarb RH, Kitson RP, Miller AH, Spencer RL, Weiss JM. The role of adrenocorticoids as modulators of immune function in health and disease: neural, endocrine and immune interactions. Brain Res Brain Res Rev. 1997 Feb;23(1-2):79-133. doi: 10.1016/s0165-0173(96)00012-4. No abstract available. PMID 9063588
- [Background] Starkman MN, Schteingart DE, Schork MA. Depressed mood and other psychiatric manifestations of Cushing's syndrome: relationship to hormone levels. Psychosom Med. 1981 Feb;43(1):3-18. doi: 10.1097/00006842-198102000-00002. PMID 6259680
- [Background] Chu JW, Matthias DF, Belanoff J, Schatzberg A, Hoffman AR, Feldman D. Successful long-term treatment of refractory Cushing's disease with high-dose mifepristone (RU 486). J Clin Endocrinol Metab. 2001 Aug;86(8):3568-73. doi: 10.1210/jcem.86.8.7740. PMID 11502780
- [Background] Carrion VG, Weems CF, Ray RD, Glaser B, Hessl D, Reiss AL. Diurnal salivary cortisol in pediatric posttraumatic stress disorder. Biol Psychiatry. 2002 Apr 1;51(7):575-82. doi: 10.1016/s0006-3223(01)01310-5. PMID 11950459
- [Background] Feder A, Coplan JD, Goetz RR, Mathew SJ, Pine DS, Dahl RE, Ryan ND, Greenwald S, Weissman MM. Twenty-four-hour cortisol secretion patterns in prepubertal children with anxiety or depressive disorders. Biol Psychiatry. 2004 Aug 1;56(3):198-204. doi: 10.1016/j.biopsych.2004.05.005. PMID 15271589
- [Background] Belanoff JK, Kalehzan M, Sund B, Fleming Ficek SK, Schatzberg AF. Cortisol activity and cognitive changes in psychotic major depression. Am J Psychiatry. 2001 Oct;158(10):1612-6. doi: 10.1176/appi.ajp.158.10.1612. PMID 11578992
- [Background] Luby JL, Heffelfinger A, Mrakotsky C, Brown K, Hessler M, Spitznagel E. Alterations in stress cortisol reactivity in depressed preschoolers relative to psychiatric and no-disorder comparison groups. Arch Gen Psychiatry. 2003 Dec;60(12):1248-55. doi: 10.1001/archpsyc.60.12.1248. PMID 14662557
- [Background] Nemeroff CB. The neurobiology of depression. Sci Am. 1998 Jun;278(6):42-9. doi: 10.1038/scientificamerican0698-42. No abstract available. PMID 9608732
- [Background] Matthews SG. Early programming of the hypothalamo-pituitary-adrenal axis. Trends Endocrinol Metab. 2002 Nov;13(9):373-80. doi: 10.1016/s1043-2760(02)00690-2. PMID 12367818
- [Background] Oitzl MS, Champagne DL, van der Veen R, de Kloet ER. Brain development under stress: hypotheses of glucocorticoid actions revisited. Neurosci Biobehav Rev. 2010 May;34(6):853-66. doi: 10.1016/j.neubiorev.2009.07.006. Epub 2009 Jul 23. PMID 19631685
- [Background] Gunnar MR, Donzella B. Social regulation of the cortisol levels in early human development. Psychoneuroendocrinology. 2002 Jan-Feb;27(1-2):199-220. doi: 10.1016/s0306-4530(01)00045-2. PMID 11750779
- [Background] Schore AN. Attachment and the regulation of the right brain. Attach Hum Dev. 2000 Apr;2(1):23-47. doi: 10.1080/146167300361309. PMID 11707891
- [Background] De Chateau P. The interaction between the infant and the environment: the importance of mother-child contact after delivery. Acta Paediatr Scand Suppl. 1988;344:21-30. doi: 10.1111/j.1651-2227.1988.tb10858.x. PMID 3067506
- [Background] Albers EM, Riksen-Walraven JM, Sweep FC, de Weerth C. Maternal behavior predicts infant cortisol recovery from a mild everyday stressor. J Child Psychol Psychiatry. 2008 Jan;49(1):97-103. doi: 10.1111/j.1469-7610.2007.01818.x. PMID 18181883
- [Background] Montgomery SM, Ehlin A, Sacker A. Breast feeding and resilience against psychosocial stress. Arch Dis Child. 2006 Dec;91(12):990-4. doi: 10.1136/adc.2006.096826. Epub 2006 Aug 3. PMID 16887859
- [Background] Taylor A, Fisk NM, Glover V. Mode of delivery and subsequent stress response. Lancet. 2000 Jan 8;355(9198):120. doi: 10.1016/S0140-6736(99)02549-0. PMID 10675176
- [Background] Essex MJ, Klein MH, Cho E, Kalin NH. Maternal stress beginning in infancy may sensitize children to later stress exposure: effects on cortisol and behavior. Biol Psychiatry. 2002 Oct 15;52(8):776-84. doi: 10.1016/s0006-3223(02)01553-6. PMID 12372649
- [Background] Koch FS, Ludvigsson J, Sepa A. Parents' psychological stress over time may affect children's cortisol at age 8. J Pediatr Psychol. 2010 Oct;35(9):950-9. doi: 10.1093/jpepsy/jsp132. Epub 2010 Jan 16. PMID 20081219
- [Background] Ainsworth MD. Patterns of infant-mother attachments: antecedents and effects on development. Bull N Y Acad Med. 1985 Nov;61(9):771-91. No abstract available. PMID 3864510
- [Background] Bartholomew K, Horowitz LM. Attachment styles among young adults: a test of a four-category model. J Pers Soc Psychol. 1991 Aug;61(2):226-44. doi: 10.1037//0022-3514.61.2.226. PMID 1920064
- [Background] Mikulincer M. Adult attachment style and individual differences in functional versus dysfunctional experiences of anger. J Pers Soc Psychol. 1998 Feb;74(2):513-24. doi: 10.1037//0022-3514.74.2.513. PMID 9491590
- [Background] Maunder RG, Hunter JJ. Attachment and psychosomatic medicine: developmental contributions to stress and disease. Psychosom Med. 2001 Jul-Aug;63(4):556-67. doi: 10.1097/00006842-200107000-00006. PMID 11485109
- [Background] Gunnar M, Quevedo K. The neurobiology of stress and development. Annu Rev Psychol. 2007;58:145-73. doi: 10.1146/annurev.psych.58.110405.085605. PMID 16903808
- [Background] Kertes DA, Donzella B, Talge NM, Garvin MC, Van Ryzin MJ, Gunnar MR. Inhibited temperament and parent emotional availability differentially predict young children's cortisol responses to novel social and nonsocial events. Dev Psychobiol. 2009 Nov;51(7):521-32. doi: 10.1002/dev.20390. PMID 19676107
- [Background] Spangler G, Grossmann KE. Biobehavioral organization in securely and insecurely attached infants. Child Dev. 1993 Oct;64(5):1439-50. doi: 10.1111/j.1467-8624.1993.tb02962.x. PMID 8222882
- [Background] Alia-Klein N, Goldstein RZ, Kriplani A, Logan J, Tomasi D, Williams B, Telang F, Shumay E, Biegon A, Craig IW, Henn F, Wang GJ, Volkow ND, Fowler JS. Brain monoamine oxidase A activity predicts trait aggression. J Neurosci. 2008 May 7;28(19):5099-104. doi: 10.1523/JNEUROSCI.0925-08.2008. PMID 18463263
- [Background] Caspi A, McClay J, Moffitt TE, Mill J, Martin J, Craig IW, Taylor A, Poulton R. Role of genotype in the cycle of violence in maltreated children. Science. 2002 Aug 2;297(5582):851-4. doi: 10.1126/science.1072290. PMID 12161658
- [Background] Jabbi M, Korf J, Kema IP, Hartman C, van der Pompe G, Minderaa RB, Ormel J, den Boer JA. Convergent genetic modulation of the endocrine stress response involves polymorphic variations of 5-HTT, COMT and MAOA. Mol Psychiatry. 2007 May;12(5):483-90. doi: 10.1038/sj.mp.4001975. Epub 2007 Mar 6. PMID 17453062
- [Background] Meyer-Lindenberg A, Buckholtz JW, Kolachana B, R Hariri A, Pezawas L, Blasi G, Wabnitz A, Honea R, Verchinski B, Callicott JH, Egan M, Mattay V, Weinberger DR. Neural mechanisms of genetic risk for impulsivity and violence in humans. Proc Natl Acad Sci U S A. 2006 Apr 18;103(16):6269-74. doi: 10.1073/pnas.0511311103. Epub 2006 Mar 28. PMID 16569698
- [Background] Ouellet-Morin I, Dionne G, Perusse D, Lupien SJ, Arseneault L, Barr RG, Tremblay RE, Boivin M. Daytime cortisol secretion in 6-month-old twins: genetic and environmental contributions as a function of early familial adversity. Biol Psychiatry. 2009 Mar 1;65(5):409-16. doi: 10.1016/j.biopsych.2008.10.003. Epub 2008 Nov 14. PMID 19013558
- [Background] Stein MB, Campbell-Sills L, Gelernter J. Genetic variation in 5HTTLPR is associated with emotional resilience. Am J Med Genet B Neuropsychiatr Genet. 2009 Oct 5;150B(7):900-6. doi: 10.1002/ajmg.b.30916. PMID 19152387
- [Background] Viding E, Frith U. Genes for susceptibility to violence lurk in the brain. Proc Natl Acad Sci U S A. 2006 Apr 18;103(16):6085-6. doi: 10.1073/pnas.0601350103. Epub 2006 Apr 10. No abstract available. PMID 16606856
- [Background] Radosevic B, Bukara-Radujkovic G, Miljkovic V, Pejicic S, Bratina N, Battelino T. The incidence of type 1 diabetes in Republic of Srpska (Bosnia and Herzegovina) and Slovenia in the period 1998-2010. Pediatr Diabetes. 2013 Jun;14(4):273-9. doi: 10.1111/j.1399-5448.2012.00898.x. Epub 2012 Aug 28. PMID 22925312
- [Background] Sepa A, Frodi A, Ludvigsson J. Could parenting stress and lack of support/confidence function as mediating mechanisms between certain environmental factors and the development of autoimmunity in children?: a study within ABIS. Ann N Y Acad Sci. 2002 Apr;958:431-5. doi: 10.1111/j.1749-6632.2002.tb03019.x. PMID 12021156
- [Background] Sepa A, Frodi A, Ludvigsson J. Mothers' experiences of serious life events increase the risk of diabetes-related autoimmunity in their children. Diabetes Care. 2005 Oct;28(10):2394-9. doi: 10.2337/diacare.28.10.2394. PMID 16186269
- [Background] Sepa A, Wahlberg J, Vaarala O, Frodi A, Ludvigsson J. Psychological stress may induce diabetes-related autoimmunity in infancy. Diabetes Care. 2005 Feb;28(2):290-5. doi: 10.2337/diacare.28.2.290. PMID 15677781
- [Background] Hagglof B, Blom L, Dahlquist G, Lonnberg G, Sahlin B. The Swedish childhood diabetes study: indications of severe psychological stress as a risk factor for type 1 (insulin-dependent) diabetes mellitus in childhood. Diabetologia. 1991 Aug;34(8):579-83. doi: 10.1007/BF00400277. PMID 1936661
- [Background] Thernlund GM, Dahlquist G, Hansson K, Ivarsson SA, Ludvigsson J, Sjoblad S, Hagglof B. Psychological stress and the onset of IDDM in children. Diabetes Care. 1995 Oct;18(10):1323-9. doi: 10.2337/diacare.18.10.1323. PMID 8721932
- [Background] Sepa A, Frodi A, Ludvigsson J. Mothers' attachment insecurity and diabetes-related autoantibodies in their infants. Ann N Y Acad Sci. 2004 Dec;1037:110-3. doi: 10.1196/annals.1337.016. PMID 15699501
- [Background] Mead VP. A new model for understanding the role of environmental factors in the origins of chronic illness: a case study of type 1 diabetes mellitus. Med Hypotheses. 2004;63(6):1035-46. doi: 10.1016/j.mehy.2004.04.014. PMID 15504572
- [Background] Target M, Fonagy P, Shmueli-Goetz Y. Attachment Representations in School-Age Children: The Development of the Child Attachment Interview (CAI). Journal of Child Psychotherapy2003;29:171-86.
- [Background] Shmueli-Goetz Y, Target M, Fonagy P, Datta A. The Child Attachment Interview: a psychometric study of reliability and discriminant validity. Dev Psychol. 2008 Jul;44(4):939-956. doi: 10.1037/0012-1649.44.4.939. PMID 18605826
- [Background] Tomori M, Rus-Makovec M. Eating behavior, depression, and self-esteem in high school students. J Adolesc Health. 2000 May;26(5):361-7. doi: 10.1016/s1054-139x(98)00042-1. PMID 10775829
- [Background] Abidin RR. Parenting stress index. Professional manual. Third ed. Lutz: PAR; 1995.
- [Background] Achenbach TM, Becker A, Dopfner M, Heiervang E, Roessner V, Steinhausen HC, Rothenberger A. Multicultural assessment of child and adolescent psychopathology with ASEBA and SDQ instruments: research findings, applications, and future directions. J Child Psychol Psychiatry. 2008 Mar;49(3):251-75. doi: 10.1111/j.1469-7610.2007.01867.x. PMID 18333930
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] Fraley RC, Waller NG, Brennan KA. An item response theory analysis of self-report measures of adult attachment. J Pers Soc Psychol. 2000 Feb;78(2):350-65. doi: 10.1037//0022-3514.78.2.350. PMID 10707340
- [Background] Collier DA, Stober G, Li T, Heils A, Catalano M, Di Bella D, Arranz MJ, Murray RM, Vallada HP, Bengel D, Muller CR, Roberts GW, Smeraldi E, Kirov G, Sham P, Lesch KP. A novel functional polymorphism within the promoter of the serotonin transporter gene: possible role in susceptibility to affective disorders. Mol Psychiatry. 1996 Dec;1(6):453-60. PMID 9154246
- [Background] Stein MB, Schork NJ, Gelernter J. Gene-by-environment (serotonin transporter and childhood maltreatment) interaction for anxiety sensitivity, an intermediate phenotype for anxiety disorders. Neuropsychopharmacology. 2008 Jan;33(2):312-9. doi: 10.1038/sj.npp.1301422. Epub 2007 Apr 25. PMID 17460615
- [Background] Philibert RA, Gunter TD, Beach SR, Brody GH, Madan A. MAOA methylation is associated with nicotine and alcohol dependence in women. Am J Med Genet B Neuropsychiatr Genet. 2008 Jul 5;147B(5):565-70. doi: 10.1002/ajmg.b.30778. PMID 18454435
- [Background] Hotamisligil GS, Breakefield XO. Human monoamine oxidase A gene determines levels of enzyme activity. Am J Hum Genet. 1991 Aug;49(2):383-92. PMID 1678250
- [Background] Frazzetto G, Di Lorenzo G, Carola V, Proietti L, Sokolowska E, Siracusano A, Gross C, Troisi A. Early trauma and increased risk for physical aggression during adulthood: the moderating role of MAOA genotype. PLoS One. 2007 May 30;2(5):e486. doi: 10.1371/journal.pone.0000486. PMID 17534436
- [Background] Nunes SF, Figueiredo IV, Pereira JS, de Lemos ET, Reis F, Teixeira F, Caramona MM. Monoamine oxidase and semicarbazide-sensitive amine oxidase kinetic analysis in mesenteric arteries of patients with type 2 diabetes. Physiol Res. 2011;60(2):309-15. doi: 10.33549/physiolres.931982. Epub 2010 Nov 29. PMID 21114364
- [Background] Wochnik GM, Ruegg J, Abel GA, Schmidt U, Holsboer F, Rein T. FK506-binding proteins 51 and 52 differentially regulate dynein interaction and nuclear translocation of the glucocorticoid receptor in mammalian cells. J Biol Chem. 2005 Feb 11;280(6):4609-16. doi: 10.1074/jbc.M407498200. Epub 2004 Dec 9. PMID 15591061
- [Background] Amstadter AB, Nugent NR, Yang BZ, Miller A, Siburian R, Moorjani P, Haddad S, Basu A, Fagerness J, Saxe G, Smoller JW, Koenen KC. Corticotrophin-releasing hormone type 1 receptor gene (CRHR1) variants predict posttraumatic stress disorder onset and course in pediatric injury patients. Dis Markers. 2011;30(2-3):89-99. doi: 10.3233/DMA-2011-0761. PMID 21508513
- [Background] Lekman M, Laje G, Charney D, Rush AJ, Wilson AF, Sorant AJ, Lipsky R, Wisniewski SR, Manji H, McMahon FJ, Paddock S. The FKBP5-gene in depression and treatment response--an association study in the Sequenced Treatment Alternatives to Relieve Depression (STAR*D) Cohort. Biol Psychiatry. 2008 Jun 15;63(12):1103-10. doi: 10.1016/j.biopsych.2007.10.026. Epub 2008 Jan 11. PMID 18191112
- [Background] Lee RS, Tamashiro KL, Yang X, Purcell RH, Harvey A, Willour VL, Huo Y, Rongione M, Wand GS, Potash JB. Chronic corticosterone exposure increases expression and decreases deoxyribonucleic acid methylation of Fkbp5 in mice. Endocrinology. 2010 Sep;151(9):4332-43. doi: 10.1210/en.2010-0225. Epub 2010 Jul 28. PMID 20668026
- [Background] Radobuljac MD, Bratina NU, Battelino T, Tomori M. Lifetime prevalence of suicidal and self-injurious behaviors in a representative cohort of Slovenian adolescents with type 1 diabetes. Pediatr Diabetes. 2009 Nov;10(7):424-31. doi: 10.1111/j.1399-5448.2009.00501.x. Epub 2009 Apr 8. PMID 19490494
- [Background] Drobnic Radobuljac M, Shmueli-Goetz Y. Attachment to Caregivers and Type 1 Diabetes in Children. Zdr Varst. 2015 Mar 13;54(2):126-30. doi: 10.1515/sjph-2015-0019. eCollection 2015 Jun. PMID 27646919